CLINICAL TRIAL: NCT06070077
Title: Enhancing Safety on the Edge: A Comprehensive Case Report on the Quality of CPR Performance in Via Ferrata Rescues
Brief Title: CPR Quality in Via Ferrata Rescues
Status: Completed | Type: Observational
Sponsor: Zdravotnicka Zachranna Sluzba Karlovarskeho Kraje, P.O. (Other)
Collaborators: Fire and Rescue Service of the Central Bohemian Region, Czech Republic (Unknown); SnT Plus, Prague, Czech Republic (Unknown)
Responsible Party: Principal Investigator, David Peran, PhD, FERC, Deputy director for quality management and scientific activities, Zdravotnicka Zachranna Sluzba Karlovarskeho Kraje, P.O.
Other Study IDs: ZZSKVK-01-2023
Record Dates: First submitted 2023-09-29; First posted 2023-10-06 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Resuscitation; Prehospital Emergency
Keywords: resuscitation; via ferrata; head up CPR; mountain CPR; quality of resuscitation
MeSH Terms: interventions — Chest Wall Oscillation; Cardiopulmonary Resuscitation

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- On ground CPR: Quality of CPR provided on the ground in a standard environment. (n=6)
  Interventions: Procedure: Chest compressions
- Via ferrata CPR: Quality of CPR provided on the via ferrata place. (n=6)
  Interventions: Procedure: Chest compressions

INTERVENTIONS:
Procedure: Chest compressions — 2 minutes of chest compressions
  Other Names: CPR

SUMMARY:
This study evaluates the effectiveness of CPR during via ferrata rescues, focusing on response quality and outcomes in challenging outdoor settings.

DETAILED DESCRIPTION:
This study investigates the quality of Cardiopulmonary Resuscitation (CPR) provided during via ferrata rescues, where challenging terrain pose unique challenges to lifesaving efforts. Via ferratas are popular adventure routes that often require swift emergency responses in cases of cardiac events or accidents. Our comprehensive case report scrutinizes CPR performance in these high-risk settings, examining critical factors such as compressions quality, rescue team coordination and safety. By shedding light on the effectiveness of CPR in via ferrata scenarios, this research aims to improve safety protocols and enhance the chances of survival for adventurers facing cardiac emergencies in remote and demanding environments.

ELIGIBILITY:
Inclusion Criteria:

* professional provider of first aid (e. g. paramedic, fire fighter, physician)
* healthy provider (e. g. no active healthcare problem that can compromise the quality of CPR)

Exclusion Criteria:

* active health care problem (e. g. fever, cough, cold etc.)
* inability to provide safety on via ferrata

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The population is formed by healthy professional providers of first aid - paramedics, fire fighters, physicians - with duty to respond.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2023-10-03 (Actual); Primary Completion 2023-10-10 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Depth of chest compressions (cm) | 2 minutes
  Quality of chest compressions in the sense of depth (5-6 cm)
Chest recoil (cm) | 2 minutes
  The quality of chest compressions in the sense of chest recoil (maximum recoil)
Frequency of chest compressions (n/min) | 2 minutes
  The quality of chest compressions in the sense of frequency (100-120 per minute)

SECONDARY OUTCOMES:
Safety of the rescuer (YES/NO) | 2 minutes
  Securing safety of the rescuer when providing CPR on via ferrata - occurrence of risk of fall

CONTACTS AND LOCATIONS:
Overall Officials: David Peran, PhD, FERC, Study Chair — Emergency Medical Services of Karlovy Vary Region; Department of Anaesthesia and Intensive Care Medicine, Third Faculty of Medicine, Charles University and FNKV University Hospital, Prague, Czech Republic; Roman Sykora, MD, PhD, Study Director — Emergency Medical Services of Karlovy Vary Region; Department of Anaesthesia and Intensive Care Medicine, Third Faculty of Medicine, Charles University and FNKV University Hospital, Prague, Czech Republic; Jana Kubalova, MD, Principal Investigator — Emergency Medical Services of Zlin Region; Czech Society for Mountain Medicine; Martin Vondra, plk. Ing., Principal Investigator — Fire and Rescue Services of Central Bohemian Region
Locations (1):
- Via Ferrata Slany, Slaný, Czech Republic, Czechia

IPD SHARING:
Plan to Share IPD: Undecided